CLINICAL TRIAL: NCT00622882
Title: Early Infectious Disease Consultation for Better Outcomes From Staphylococcus Aureus Bacteremia
Brief Title: Early Infectious Disease Consultations in Staphylococcus Aureus Bacteremia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Medicine, Professor Paul Ananth Tambyah, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DSRB-B/06/274; DSRB-B/06/274
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Staphylococcus Aureus Bacteremia
Keywords: Staphylococcus aureus; Bacteremia; Outcome; Mortality; Recurrence; Infectious Diseases specialists
MeSH Terms: conditions — Staphylococcal Infections; Bacteremia; Recurrence | interventions — Health Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ID (Active Comparator): Patients receiving an early Infectious disease consultation ( within first 48 hours of a positive blood culture)
  Interventions: Other: infectious disease specialist consultation
- NO ID (No Intervention): Includes those patients who do not receive an Infectious disease consultation in the first 48 hours

INTERVENTIONS:
Other: infectious disease specialist consultation — Randomised trial to determine the utility of an early Infectious disease Consultation in Staphylococcus aureus bacteremic patients ( in the first 48 hours of a positive blood culture)
  Other Names: Health Services
  Arms: ID

SUMMARY:
The primary objective is to determine if early infectious disease (ID) consultation (defined as within 48 hours of a positive blood culture) will reduce mortality rates from Staphylococcus aureus bacteremia (SAB). This study will also determine if such consultations could reduce the duration of hospitalisation, recurrence and financial costs in patients with this infection.

DETAILED DESCRIPTION:
Bacteremia is a serious manifestation of Staphylococcus aureus infection with an attributable mortality as high as 25% in MRSA bacteremia. More than a third of patients end up with complications such as endocarditis, osteomyelitis or pneumonia.

Overall the outcome of patients with respect to mortality or recurrence is better in patients who have an eradicable focus and have received an appropriate antibiotic dose and duration. Also complicated bacteremia is more common in patients with

* persistent bacteremia or fever
* prosthetic device
* new murmur
* skin findings of a systemic infection

Based on this evidence, an ID consultation could improve the outcomes of patients with SAB by

* Advising adequate antibiotic dosage and duration
* Sourcing out and counselling eradication of any focus of infection

ELIGIBILITY:
Inclusion Criteria:

* All inpatients at the National University Hospital with Staphylococcus aureus (both methicillin sensitive and methicillin resistant) bacteremia isolated within the defined time period

Exclusion Criteria:

* Patients who died or were discharged before the notification from the laboratory
* Neonates
* Polymicrobial bacteremia

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
mortality | 1 year

SECONDARY OUTCOMES:
recurrence | 2 year
duration of hospitalisation | 1 year
financial costs of hospitalisation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Tambyah, MD, Principal Investigator — National University of Singapore
Locations (1):
- National University Hospital, Singapore, Singapore